CLINICAL TRIAL: NCT00089999
Title: A Phase II, Open-Label, Randomized, Parallel-Group Multicenter Trial Comparing Two Schedules of GW572016 as First-Line Monotherapy in Patients With Advanced or Metastatic Breast Cancer
Brief Title: Lapatinib In Chemotherapy-Naive Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF20009
Record Dates: First submitted 2004-08-18; First posted 2004-08-23 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Neoplasms, Breast
Keywords: lapatinib; advanced; metastatic breast cancer; GW572016; ErbB2
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lapatinib

SUMMARY:
This phase II study will evaluate and compare the efficacy and tolerability of two dose schedules (1500 mg QD and 500 mg BID) of oral Lapatinib as treatment for patients with advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed invasive breast cancer with incurable stage IIIB, IIIC with T4 lesion or stage IV disease at primary diagnosis or at relapse after curative intent surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Documented amplification of ErbB2 by Fluorescence in situ hybridization (FISH)
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST)
* Adequate renal, hepatic and cardiac function

Exclusion criteria:

* Prior chemotherapy, immunotherapy, biologic therapy or anti-ErbB1/ErbB2 therapy other than adjuvant therapy. [Prior neo-adjuvant or adjuvant therapy (including trastuzumab) will be allowed provided it was stopped at least 12 months before study entry.
* Patients with active brain metastases
* Patients with bilateral breast cancer, bone metastases as the only disease site or metastases to more than 30% of the hepatic parenchyma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- GSK Investigational Site, Hollywood, Florida, United States
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, Pokfulam, Hong Kong
- India (3):
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, Pune
- Malaysia (3):
  - GSK Investigational Site, Bandar Tun Razak, Cheras
  - GSK Investigational Site, Kubang Kerian
  - GSK Investigational Site, Tanjong Bungah
- Mexico (3):
  - GSK Investigational Site, Ixtaltepec / Espinal, Oaxaca
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, México
- Pakistan (3):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
  - GSK Investigational Site, Rawalpindi
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao
- Poland (3):
  - GSK Investigational Site, Bydogoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Taipei, Taiwan

REFERENCES:
- [Background] Lipton A, Leitzel K, Ali SM, Carney W, Platek G, Steplewski K, Westlund R, Gagnon R, Martin AM, Maltzman J. Human epidermal growth factor receptor 2 (HER2) extracellular domain levels are associated with progression-free survival in patients with HER2-positive metastatic breast cancer receiving lapatinib monotherapy. Cancer. 2011 Nov 1;117(21):5013-20. doi: 10.1002/cncr.26101. Epub 2011 Mar 31. PMID 21456017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) with histologically confirmed invasive breast cancer with incurable stage IIIb, stage IIIc with T4 lesion, or stage IV disease at primary diagnosis or at relapse after curative-intent surgery and whose tumors overexpressed ErbB2 protein, documented by FISH were eligible for inclusion in this phase II study.
Groups:
- Lapatinib 1500 mg QD: Participants received lapatinib 1500 milligram (mg) orally once daily (QD). Treatment was continued for 12 weeks or until disease progression or withdrawal from treatment for another reason. After Week 12, participants with clinical benefit had the option to continue with the lapatinib therapy at the same dose and schedule, until disease progression, provided the treatment was tolerated.
- Lapatinib 500 mg BID: Participants received lapatinib 500 mg orally twice daily (BID). Treatment was continued for 12 weeks or until disease progression or withdrawal from treatment for another reason. After Week 12, participants with clinical benefit had the option to continue with the lapatinib therapy at the same dose and schedule, until disease progression, provided the treatment was tolerated.
Period: Overall Study
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Started | 69 | 69
Completed | 0 | 0
Not Completed | 69 | 69
Not completed — Adverse Event | 4 | 7
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Radiological Progression of Cancer | 52 | 44
Not completed — Symptomatic Progression of Cancer | 2 | 5
Not completed — Death | 3 | 3
Not completed — Poor General Condition | 1 | 0
Not completed — Clinical Progression | 1 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Patient Underwent Surgery | 2 | 0
Not completed — Skin Nodule Over Right Mastectomy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lapatinib 1500 mg QD: Participants received lapatinib 1500 mg orally QD. Treatment was continued for 12 weeks or until disease progression or withdrawal from treatment for another reason. After Week 12, participants with clinical benefit had the option to continue with the lapatinib therapy at the same dose and schedule, until disease progression, provided the treatment was tolerated.
- Lapatinib 500 mg BID: Participants received lapatinib 500 mg orally BID. Treatment was continued for 12 weeks or until disease progression or withdrawal from treatment for another reason. After Week 12, participants with clinical benefit had the option to continue with the lapatinib therapy at the same dose and schedule, until disease progression, provided the treatment was tolerated.
- Total: Total of all reporting groups
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (14.27) | 53.4 (13.66) | 53.3 (13.92)
Gender [Count of Participants; unit: Participants]
  Female | 69 | 69 | 138
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2 | 1 | 3
  Black | 0 | 1 | 1
  Asian | 36 | 35 | 71
  American Hispanic | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Best Overall Response (OR) of Confirmed Complete Response (CR) or Partial Response (PR), as Assessed by the Independent Review Committee (IRC)
Description: OR is defined as the number of participants achieving either a confirmed CR or PR, per Response Evaluation Criteria in Solid Tumors (RECIST, v 1.0). Best OR is defined as the best response recorded from the start of treatment until progressive disease (PD)/recurrence. CR is defined as the disappearance of all target lesions (TLs) and non-TLs. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s), as assessed by the IRC. PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of >= 1 new lesions or unequivocal progression of existing non-TLs. Responses were confirmed at subsequent assessments made >=28 days after the original response. Participants with an unknown or missing response are treated as non-responders.
Time Frame: From the date of the first dose of investigational product to the first documented evidence of a confirmed CR or PR (up to Study Week 103)
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Participants
  CR | 0 | 0
  PR | 15 | 18
Statistical Analysis 1: Comparison: Lapatinib 1500 mg QD vs Lapatinib 500 mg BID; Test type: Superiority or Other; p = 0.691, Fisher Exact; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.3 to 1.9]

2. Primary Outcome: Number of Participants With a Best Overall Response (OR) of Confirmed Complete Response (CR) or Partial Response (PR), as Assessed by the Investigator
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Participants
  CR | 1 | 2
  PR | 16 | 20
Statistical Analysis 1: Comparison: Lapatinib 1500 mg QD vs Lapatinib 500 mg BID; Test type: Superiority or Other; p = 0.443, Fisher Exact; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 1.6] — Overall Response (i.e. sum of Complete and Partial Responses) comparison

3. Secondary Outcome: Percentage of Participants With Clinical Benefit (CR or PR or Stable Disease [SD] for at Least 24 Weeks), as Assessed by the IRC and Investigator
Description: Clinical benefit is defined as the numer of participants achieving either a confirmed CR (disappearance of all target lesions (TLs) and non-TLs) or PR (at least a 30% decrease in the sum of the longest diameters (LD) of TLs, taking as a reference the Baseline sum LD and no PD,or complete resolution of TLs and the persistence of one or more non-TLs)or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [at least a 20% increase in the sum of the LD of target lesions, taking as a reference, the smallest sum LD recorded since the treatment started or the appearance of 1 or more new TLs or non-TLs and/or unequivocal progressionn of existing non-target lesions], taking as reference, the smallest sum LD since the treatment started) for at least 24 weeks. This was based on confirmed responses from the investigator assessment of clinical benefit.
Time Frame: From the date of the first dose of investigational product until the date of disease progression or death due to breast cancer (up to Study Week 103)
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Groups:
- Lapatinib 1500 mg QD: Participants received lapatinib 1500 mg orally QD. Treatment was continued for 12 weeks or until disease progression or withdrawal from treatment for another reason. After Week 12, participants with clinical benefit had the option to continue with the lapatinib therapy at the same dose and schedule, until disease progression, provided the treatment was tolerated.Participants received lapatinib 1500 mg orally QD. Treatment was continued for 12 weeks or until disease progression or withdrawal from treatment for another reason. After Week 12, participants with clinical benefit had the option to continue with the lapatinib therapy at the same dose and schedule, until disease progression, provided the treatment was tolerated.
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Percentage of Participants
  IRC | 29.0 | 33.3
  Investigator | 29.0 | 40.6

4. Secondary Outcome: Time to Response, as Assessed by the IRC and Investigator
Description: Time to response is defined as the time from randomization until the first documented evidence of a PR or CR (whichever status is recorded first). Analysis was based on responses confirmed at a repeat assessment made at least 4 weeks after the initial response, with the time to response taken as the first time the response was observed, not the confirmation assessment. Participants who withdraw with no tumor response were censored at the date of withdrawal from the study. CR is defined as the disappearance of all TLs and non-TLs. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of one or more non-TL(s). PD is defined as at least a 20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-TLs.
Time Frame: From the date of the first dose of investigational product until the first documented evidence of a PR or CR (up to Study Week 103)
Population: ITT Population. Only those participants with CR or PR were analyzed (represented by n=X in the category titles). Different participants may have been analyzed by the IRC and the Investigator, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Weeks
  IRC, n=15, 18 | 7.9 [7 to 12] | 7.9 [7 to 20]
  Investigator, n=17, 22 | 8.0 [7 to 19] | 8.0 [5 to 46]

5. Secondary Outcome: Duration of Response (DoR), as Assessed by the IRC and Investigator
Description: DoR is defined for the subset of par. who had a confirmed CR (disappearance of all target lesions (TLs) and non-TLs) or PR (at least a 30% decrease in the sum of the longest diameters (LD) of TLs, taking as a reference the Baseline sum LD and no PD, or complete resolution of TLs and the persistence of >= 1 non-TL[s]) as the time from the first documented evidence of a CR or PR until the first documentation of radiological PD or death due to breast cancer, if sooner. PD is defined as >=20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of >= 1 new lesions or unequivocal progression of existing non-TLs. For par. who did not progress or die, DoR was censored on the date of the last radiological scan. If a par.had only a Baseline visit or did not have a date of a radiological scan that was later than the date of initiation of anti-cancer therapy, DoR was censored at the start date of treatment.
Time Frame: From the first documented evidence of a PR or CR until the earlier of the date of disease progression or the date of death due to breast cancer (up to Study Week 103)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Weeks
  IRC,n=15, 18 | 27.6 [20.1 to 39.4] | 29.0 [20.3 to NA] — The upper limit of the 95% confidence interval could not be determined (not reached) because there were not enough events to be able to calculate it.
  Investigator, n=17, 22 | 27.6 [15.4 to 39.4] | 29.0 [15.7 to 36.1]

6. Secondary Outcome: Progression-free Survival, as Assessed by the IRC and Investigator
Description: Progression-free survival is defined as the time from randomization until the earliest date of disease progression or death due to any cause, if sooner. Disease progression was based on the IRC's and investigator's assessments of the objective evidence (e.g., radiological scans and medical photographs). For participants who did not progress, or die, progression-free survival was censored at the time of the last IRC assessed radiological scan.
Time Frame: From the date of the first dose of investigational product until the earlier of the date of disease progression or death due to any cause (up to Study Week 103)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Weeks
  IRC | 19.6 [16.4 to 28.1] | 24.4 [19.7 to 35.9]
  Investigator | 17.6 [12.1 to 20.0] | 20.3 [13.3 to 24.4]

7. Secondary Outcome: Time to Treatment Failure, as Assessed by IRC and Investigator
Description: Time to treatment failure is calculated as the interval between the date of randomization and the occurrence of local tumor progression (including ipsilateral [on the same side] and controlateral breast tumor progression), distant tumor progression, permanent treatment discontinuation (either for the experimental or conventional treatment arm), or death due any cause. For participants who did not progress, die or discontinue early, time to treatment failure was censored at the last scan date.
Time Frame: From randomization until the first documented sign of disease progression, death due to any cause, or early discontinuation from investigational product (up to Study Week 103)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Weeks
  IRC | 15.7 [11.6 to 19.3] | 17.0 [13.1 to 20.3]
  Investigator | 12.3 [10.0 to 19.6] | 16.1 [12.3 to 23.1]

8. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations. Refer to the general AE/SAE module for a list of non-serious AEs and SAEs.
Time Frame: From the date of the first dose of investigational product until 30 days after the last dose of investigational product (up to study week 192)
Population: Safety Population: all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 69 | 69
Participants
  Any AE | 65 | 61
  Any SAE | 15 | 18

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product to 30 days after the last dose (up to Study Week 192).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of investigational product , according to the actual treatment received.
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Serious Adverse Events (participants affected / at risk) | 15/69 | 18/69
Other Adverse Events (participants affected / at risk) | 58/69 | 53/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg QD (N=69) | Lapatinib 500 mg BID (N=69)
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 1 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 2
Convulsion (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg QD (N=69) | Lapatinib 500 mg BID (N=69)
Diarrhoea (Gastrointestinal disorders) | 30 | 34
Nausea (Gastrointestinal disorders) | 10 | 9
Vomiting (Gastrointestinal disorders) | 11 | 8
Dyspepsia (Gastrointestinal disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Stomatitis (Gastrointestinal disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 23 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 18
Dry skin (Renal and urinary disorders) | 3 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Headache (Nervous system disorders) | 9 | 8
Dizziness (Nervous system disorders) | 3 | 7
Asthenia (General disorders) | 6 | 10
Pyrexia (General disorders) | 5 | 4
Alanine aminotransferase increased (Investigations) | 5 | 6
Blood alkaline phosphatase increased (Investigations) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 3 | 6
Influenza (Infections and infestations) | 6 | 6
Anorexia (Metabolism and nutrition disorders) | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.